CLINICAL TRIAL: NCT04824287
Title: The Effect of Pelvic Floor Muscle Exercises on Bowel Evacuation Problems and Quality of Life in Individuals With Closed Stoma
Brief Title: Pelvic Floor Muscle Exercises Effect After Stoma Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek Aktaş (Other)
Responsible Party: Sponsor-Investigator, Dilek Aktaş, Research Assistant Doctor, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/61
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Stoma
Keywords: stoma; stoma and wound care nurse; pelvic floor exercises; bowel evacuation problems; quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): pelvic floor exercise
  Interventions: Other: pelvic floor muscle exercise
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: pelvic floor muscle exercise — pelvic floor muscle exercises training from the researcher using the Roy Adaptation Model in addition to routine discharge training Face-to-face training was given to the individuals in the experimental group on the day before the operation, on the second and third postoperative days, and on the day of discharge. The training continued with phone calls at the first, second and third weeks and the first, second, third, and sixth months after the surgery Patients practiced exercises 6 month after surgery
  Arms: Experimental

SUMMARY:
This study was conducted to evaluate the effect of pelvic floor muscle exercises on bowel evacuation problems and quality of life in individuals after stoma closure.

DETAILED DESCRIPTION:
Sample of study was calculated as 32 using G*Power Software (ver. 3.1.9.2) for 80% power and medium effect size (f=0.25) at 95% confidence level in line with the data of Lin et al. Participants were assigned to the experimental and control groups by the stratified block randomization method. The locks were assigned to layers using Microsoft Excel.

The individuals in the experimental group received pelvic floor muscle exercises training from the researcher using the Roy Adaptation Model in addition to routine discharge training. The patients received a PFME training booklet prepared by the researcher. Face-to-face training was given to the individuals in the experimental group on the day before the operation, on the second and third postoperative days, and on the day of discharge. The training continued with phone calls at the first, second and third weeks and the first, second, third, and sixth months after the surgery. Data was collected a day before discharge, first, second, third, and sixth months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 75,
* Being literate,
* Having a stoma due to colorectal cancer,
* Having no previous anal trauma,
* Having no anal surgery other than colorectal cancer surgery,
* Having no congenital anorectal anomaly,
* Having no neurological problem,
* Having no physical disability,
* Having no previous experience of PFMEs before the surgery,
* Being cognitively able to answer questions

Exclusion Criteria:

* Wanting to leave the study,
* Having had previous biofeedback and electrical stimulation therapy applications,
* Having another stoma,
* Not being reachable by phone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Bowel Evacuation Habits | 6 month
  evaluated with "Assessment Form for Bowel Evacuation Habits and Psychosocial Problems". This form was developed by the researcher. Patients answer the question yes or no
Wexner Scale Score | 6 month
  Wexner Scale used to evaluate fecal incontinence. Minimum point is "0" an maximum point is "20". A score of 1 or above indicates a fecal incontinence problem
Psychosocial Problems | 6 month
  evaluated with "Assessment Form for Bowel Evacuation Habits and Psychosocial Problems". This form was developed by the researcher. The form include questions about psychosocial problems related bowel evacuation problems Patient answer the questions yes or no
Health-related Quality of Life | 6 month
  evaluated with Short Form 36 (SF-36) Health-related Quality of Life Scale. This scale include 8 subdimensions. scale does not have a single total score: the score for each dimension is calculated separately. For each subdimension minimum point is 0 and maximum point is 100. Higher score indicate best quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Aktaş, Principal Investigator — Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Nursing, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No